CLINICAL TRIAL: NCT06952140
Title: Hemodynamic Effects of Ketone Esters in Patients With Sepsis Induced Cardiomyopathy
Acronym: KetoSIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KetoSIC
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Sepsis Induced Cardiomyopathy
Keywords: Sepsis induced cardiomyopathy; Sepsis; Hemodynamics; Ketone ester; Ketones; Echocardiography; Randomized controlled trial; Cross-over trial; Cardiovascular
MeSH Terms: conditions — Sepsis; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: As this is a cross-over trial participants will receive both active treatment and placebo. Participants will be randomized 1:1 to receive A) active treatment followed by placebo or B) placebo followed by active treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone ester followed by placebo (Experimental)
  Interventions: Dietary Supplement: Ketone ester; Dietary Supplement: Placebo
- Placebo followed by ketone ester (Experimental)
  Interventions: Dietary Supplement: Ketone ester; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — Ketone ester: 3-hydroxybutyrate as enteral bolus (500 mg/kg)
Dietary Supplement: Placebo — Maltodextrin (isovolumic and isocaloric placebo) as enteral bolus

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection and is associated with a high mortality rate in the ICU. Sepsis induced cardiomyopathy (SICM) is a multi-factorial process that appears in approximately 50% of patients with sepsis/septic shock and is associated with increased mortality. It is suggested that ketone bodies are more efficient substrates of energy metabolism than glucose, with a lower oxygen consumption per ATP-molecule produced and that the failing human heart increases the capacity to metabolize ketones. Previous studies have found acute beneficial hemodynamic effects of ketone esters in patients with chronic heart failure and cardiogenic shock, respectively. Improved hemodynamics and reduced systemic oxygen consumption as an effect of ketone esters might be of great benefit in patients admitted to the ICU. Thus, the investigators aim to investigate the hemodynamic effects of ketone esters in patients with sepsis induced cardiomyopathy in this randomized, placebo-controlled, double-blinded, cross-over, acute intervention study. .

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age admitted to the the intensive care unit (ICU)
* LVEF < 40% determined by a screening echocardiography (two projections: apical 4 chamber and 2 chamber) and analysed according to the Simpson biplane method
* Ability for study personnel to perform transthoracic echocardiography
* Suspected or documented infection (suspected infection is defined as ongoing antibiotic treatment and/or body fluid culture sampling performed within 72 hours before screening)

Exclusion Criteria:

* Diagnosis of heart failure with reduced ejection fraction prior to ICU admission according to health records
* Surgical cause of ICU admission
* For patients in shock: Other primary causes of shock than sepsis (i.e. hypovolemia, haemorrhage, cardiogenic etiology, pulmonary embolism, anaphylaxis)
* Blood pH < 7.20
* Severe gastroparesis
* Inability to position a nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Global longitudinal strain | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
  Echocardiographic measure obtained from transthoracic echocardiography

SECONDARY OUTCOMES:
Left ventricular ejection fraction | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
  Echocardiographic measure obtained from transthoracic echocardiography
Mean arterial pressure | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
  Obtained from invasive blood pressure measurement (arterial line)
Cardiac output | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
  Obtained from transthoracic echocardiography
Peripheral blood oxygen saturation | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
Arterial blood pH | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
Arterial blood lactate | From intervention to 3 hours after intervention (this is assessed for both treatment arms)
Accumulated norepinephrine | From intervention to 3 hours after intervention (this is assessed for both treatment arms)

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MPH, MSc, PhD, Principal Investigator — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte